CLINICAL TRIAL: NCT01991184
Title: An Open-Label, Phase I, Dose-Escalation Study Evaluating The Safety And Tolerability Of Gdc-0853 In Patients With Relapsed Or Refractory B-Cell Non-Hodgkin's Lymphoma And Chronic Lymphocytic Leukemia
Brief Title: A Study of GDC-0853 in Patients With Resistant B-Cell Lymphoma or Chronic Lymphocytic Leukemia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO29089
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Lymphocytic Leukemia, Chronic, Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphoid; Bronchiolitis Obliterans Syndrome; Lymphoma, Large B-Cell, Diffuse | interventions — fenebrutinib

ARMS (1):
- Dose-escalation (Experimental)
  Interventions: Drug: GDC-0853

INTERVENTIONS:
Drug: GDC-0853 — Multiple escalating doses
  Other Names: Fenebrutinib

SUMMARY:
This open-label, Phase I study will evaluate the safety, tolerability, and pharmacokinetics of increasing doses of GDC-0853 in patients with relapsed or refractory B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia. In a dose-expansion part, GDC-0853 will be assessed in subsets of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* ECOG score of 0-1
* One of the following histologically-documented hematologic malignancies for which no effective standard therapy exists: indolent non Hodgkin's lymphoma (NHL), follicular lymphoma (FL), diffuse large B-cell lymphoma (DLBCL), mantle cell lymphoma (MCL), or chronic lymphocytic leukemia (CLL)
* At least one site of disease that, as seen on CT scan, is > 1.5 cm in the greatest transverse diameter or > 1.0 cm in short axis diameter (except for patients with CLL)
* An available tumor specimen
* Adequate hematologic and organ function
* For female patients of childbearing potential and male patients with partners of childbearing potential, use of effective contraceptive(s) as defined by protocol for the duration of the study

Exclusion Criteria:

* Life expectancy < 12 weeks
* < 3 weeks since the last anti-tumor therapy, including chemotherapy, biologic, experimental, hormonal or radiotherapy (with the exception of leuprolide or similar medications for prostate cancer)
* Recent major surgical procedure or traumatic injury, or unhealed incisions or wounds
* Active infection requiring IV antibiotics
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
* Primary CNS malignancy or untreated/active CNS metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control)
* History of other malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin cancer, Stage I uterine cancer, or other cancers with a similar outcome
* Cardiovascular dysfunction, including ventricular dysrhythmias or risk factors for ventricular dysrhythmias
* Pregnancy, or lactation
* Any other diseases that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of dose-limiting toxicities (DLTs) of GDC-0853 | Approximately 1 year
Safety: Maximum tolerated dose (MTD) of GDC-0853 | Approximately 1 year

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | Approximately 2 years
Pharmacokinetics: Area under the concentration-time curve (AUC) of GDC-0853 | 35 days
Pharmacokinetics: Maximum concentration (Cmax) of GDC-0853 | 35 days
Objective response to GDC-0853 | Approximately 2 years
Progression-free survival | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (10):
- United States (7):
  - Stanford Cancer Center, Stanford, California
  - Washington University School of Medicine, St Louis, Missouri
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Willamette Valley Cancer Ctr - 520 Country Club, Eugene, Oregon
  - Oregon Health Sciences Uni, Portland, Oregon
  - Sarah Cannon Cancer Center - Tennessee Oncology, Pllc, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (3):
  - Princess Alexandra Hospital Woolloongabba; Clinical Hematology and Medical Oncology, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre; Department of Haematology, Melbourne, Victoria
  - Linear Clinical Research Limited, Nedlands, Western Australia